CLINICAL TRIAL: NCT02012712
Title: Personal Health Records and Elder Medication Use Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Elizabeth A Chrischilles, Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 200708714; R18HS017034 (AHRQ)
Record Dates: First submitted 2013-11-06; First posted 2013-12-16 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2017-03

CONDITIONS: Adverse Reaction to Drug; Health Behavior; Medication Adherence; Physician-Patient Relations
Keywords: Personal health record; medication management; patient safety
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Health Behavior; Medication Adherence | interventions — Health Records, Personal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Personal Health Record (PHR) (Experimental): Subjects were sent an invitation to use an online Personal Health Record (PHR)
  Interventions: Behavioral: Personal Health Record (PHR)
- Usual care (No Intervention): Subjects received usual care (no invitation or access to the study PHR)

INTERVENTIONS:
Behavioral: Personal Health Record (PHR) — Iowa PHR is a Web-based application that features a tabbed interface design. Users can enter, view, and print their current and past medicines, allergies, health conditions, and health event tracking over time. An embedded tutorial video provides assistance with the system. The PHR was developed and refined using participatory design and focus group sessions as well as evaluation in a usability laboratory. The resulting design emphasizes the reduction of physical and cognitive demands on users, focusing on simplicity, readability, and quick navigation.
  Iowa PHR displayed a message when a user entered a medication with an associated Assessing Care of Vulnerable Elders project (ACOVE-3) safety concern. This included 16 safety issues for 12 drugs or drug classes with safety concerns. We also adapted four general medication use patient safety indicators from the ACOVE project and displayed them to all users on a rotating basis upon login.
  Arms: Personal Health Record (PHR)

SUMMARY:
Purpose: To examine the impact of a personal health record (PHR) on medication use safety among older adults.

Background: Online PHRs have potential as tools to manage health information. We know little about how to make PHRs accessible for older adults and what effects this will have.

Methods: A PHR was designed and pretested with older adults and tested in a six-month randomized controlled trial. After completing mailed baseline questionnaires, eligible computer users aged 65 and over were randomized 3:1 to be given access to a PHR (n=802) or serve as a standard care control group (n=273). Follow-up questionnaires measured change from baseline medication use, medication reconciliation behaviors, and medication management problems.

ELIGIBILITY:
Inclusion Criteria:

* Computer use within the past month.
* Age 65+

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1163 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Mean (SD) number of prescription drugs | Baseline and 6 months
Mean (SD) number of over-the-counter drugs | Baseline and 6 months
Any change in medication use in past 3 months | Baseline and 6 months
Started prescription drug | Baseline and 6 months
Stopped prescription drug | Baseline and 6 months
Changed strength/dose of prescription drug | Baseline and 6 months
Keep list of current medications | Baseline and 6 months
Reason for medications on list | Baseline and 6 months
Usually shows medication list to doctor | Baseline and 6 months
Put over-the-counter drugs on list | Baseline and 6 months
Updated list in past 3 months | Baseline and 6 months
At last doctor visit, asked whether keep a medication list | Baseline and 6 months
At last doctor visit, had medication list | Baseline and 6 months
At last doctor visit showed medication list | Baseline and 6 months
Someone asked about medication strength at last doctor visit (for all medications) | Baseline and 6 months
Someone asked about medication strength at last doctor visit (for some medications) | Baseline and 6 months
At last doctor visit, doctor compared records with what patient said they were taking | Baseline and 6 months
At last doctor visit, differences found between doctor and patient medication records | Baseline and 6 months
Use of potentially inappropriate medications (ACOVE) | Baseline and 6 months
  List of potentially inappropriate medications derived from the Assessing Care of Vulnerable Elders project (ACOVE-3)
  Shrank WH, Polinski JM, Avorn J. Quality Indicators for Medication Use in Vulnerable Elders. J Am Geriatr Soc 2007;55:S373-S382.
Taking 2 or more NSAIDS (including aspirin) | Baseline and 6 months
Mean (SD) number of medication management problems | Baseline and 6 months
Knows how to recognize side effects | 6 months
Medication side effects in past 3 months | Baseline and 6 months
Mean (SD) modified Morisky adherence score | Baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Chrischilles, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Background] Hourcade, J.P., Chrischilles, E.A., Gryzlak, B.M., Hanson, B.M., Dunbar, D.E., Eichmann, D.A. and Lorentzen, R.R. (2011). Design Lessons for Older Adult Personal Health Records Software from Older Adults. Proceedings of 6th International Conference on Universal Access in Human-Computer Interaction, held as part of HCI International. Lecture Notes in Computer Science, 6766, 176-85.
- [Background] Witry MJ, Doucette WR, Daly JM, Levy BT, Chrischilles EA. Family physician perceptions of personal health records. Perspect Health Inf Manag. 2010 Jan 1;7(Winter):1d. PMID 20697465
- [Result] Chrischilles EA, Hourcade JP, Doucette W, Eichmann D, Gryzlak B, Lorentzen R, Wright K, Letuchy E, Mueller M, Farris K, Levy B. Personal health records: a randomized trial of effects on elder medication safety. J Am Med Inform Assoc. 2014 Jul-Aug;21(4):679-86. doi: 10.1136/amiajnl-2013-002284. Epub 2013 Dec 10. PMID 24326536
- See also: [Manuscript] Design Lessons for Older Adult Personal Health Records Software from Older Adults — http://link.springer.com/chapter/10.1007%2F978-3-642-21663-3_19
- See also: Project final report — http://healthit.ahrq.gov/ahrq-funded-projects/personal-health-records-and-elder-medication-use-quality